CLINICAL TRIAL: NCT01734018
Title: A Multicenter, Prospective, Non-Interventional Study Evaluating Response Parameters During and After Therapy With PEGASYS (Peginterferon Alfa-2a 40KD) in Subjects With HBeAg Positive or HBeAg Negative Chronic Hepatitis B
Brief Title: An Observational Study of Pegasys (Peginterferon Alfa-2a) in Patients With HBeAg-Positive or HBeAg-Negative Chronic Hepatitis B
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25614
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, prospective, observational study will evaluate the efficacy and safety of Pegasys (peginterferon alfa-2a) in routine clinical practice in patients with HBeAg-positive or HBeAg-negative chronic hepatitis B. Eligible patients receiving treatment with Pegasys according to standard of care and the summary od product characteristics/local labelling will be followed for the duration of treatment and up to 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* HBeAg-positive or HBeAg-negative serologically proven chronic hepatitis B with or without cirrhosis
* Elevated serum ALT > ULN (upper limit of normal) but </=10 x ULN according to local label

Exclusion Criteria:

* Contra-indications to Pegasys as detailed in the label
* Co-infection with hepatitis A, hepatitis B or HIV
* Concomitant therapy with telbivudine (concomitant peginterferon alfa-2a therapy is contra-indicated according to telbivudine label)
* Pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis B receiving treatment with Pegasys
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in HBsAg (IU/ml) levels during therapy (up to 48 weeks) and follow-up | from baseline to up to approximately 3 years
Change in HBV DNA (IU/ml) during therapy (up to 48 weeks) and follow-up | from baseline to up to approximately 3 years

SECONDARY OUTCOMES:
Percentage of patients with sustained immune control (sustained HBV DNA <2000 IU/ml in HBeAg-negative and HBeAg-positive patients or HBeAg seroconversion in HBeAg-positive patients) | approximately 4 years
Percentage of patients with normalisation of serum alanine transaminase (ALT) levels | approximately 4 years
Percentage of patients with HBsAg clearance/seroconversion | approximately 4 years
Safety: Incidence of adverse events | approximately 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Germany (2):
  - Berlin
  - Leipzig